CLINICAL TRIAL: NCT06974708
Title: Interactive Virtual Occupational Safety Training Designed With and for Ohio Home Healthcare Workers and Agencies
Brief Title: Interactive Virtual Occupational Safety Training Designed for Home Healthcare Workers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Kansas Medical Center (Other); Virginia Commonwealth University (Other)
Responsible Party: Principal Investigator, Carolyn Sommerich, Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 240315-036; WSIC25-240315-036 (Other Grant/Funding Number: BWC Workforce Safety Innovation Center)
Record Dates: First submitted 2025-04-24; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Learning
Keywords: home healthcare; training; occupational safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot study of generalizability of the enhanced Home Healthcare Virtual Simulation Training System (Experimental)
  Interventions: Other: Home Healthcare Virtual Simulation Training System

INTERVENTIONS:
Other: Home Healthcare Virtual Simulation Training System — Interactive Virtual Occupational Safety Training Software Program for Home Healthcare Workers and Agencies

SUMMARY:
Overview. The investigators will collect preliminary data on the extent to which the knowledge gained from the enhanced HH-VSTS transfers to a real-world environment. Following abbreviated use of the enhanced HH-VSTS, participants will perform a walk-through of a realistic environment to assess their learning.

DETAILED DESCRIPTION:
The pilot test will use a quasi-experimental design with between groups and within subjects features to evaluate the generalizability of the enhanced HH-VSTS to a home setting. Participants will complete one of the three training modules in the HH-VSTS and then perform an actual walk-through of a simulated home setting during which they will be asked to identify any hazard that they think they recognize. The simulated home setting is a furnished apartment in Atwell Hall that is used for training OT and PT students. The primary outcome is Learning Transfer, assessed by hazard identification. The secondary outcome is the hazard response.

ELIGIBILITY:
Inclusion Criteria:

* have no formal training in home safety, and
* ≥18 years old, and
* able to read and write in English.

Exclusion Criteria:

* Participant in a prior study about home healthcare worker occupational safety training
* Individuals who meet criteria for Pre-existing Conditions Related to Cybersickness (a set of 4 screening questions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Learning transfer as measured by hazard identification | immediately after exposure to the intervention
  Number of hazards identified in the environment

SECONDARY OUTCOMES:
Hazard Response | immediately after exposure to the intervention
  Response consists of what participant would do about identified hazard and how they would talk with client/family about the hazard and how to address it. Hazard response will be defined using a coding scheme that we developed previously (REF). The coding scheme includes three response categories: (1) Optimal, which is an effective response without negative impact to either the home healthcare worker (HHW) or care recipient; (2) Mixed, defined as a response that can reduce the hazard, but can negatively impact either the HHW or the care recipient; and (3) Suboptimal, in which the hazard response is ineffective or inappropriate.
  REF: This is the publication we reference for this measurement: Wills CE, Polivka BJ, Darragh A, Lavender S, Sommerich C, Stredney D. "Making Do" decisions: How home healthcare personnel manage their exposure to home hazards. Western Journal of Nursing Research. 2016;38(4):411-426

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Darragh AR, Lavender S, Polivka B, Sommerich CM, Wills CE, Hittle BA, Chen R, Stredney DL. Gaming Simulation as Health and Safety Training for Home Healthcare Workers. Clin Simul Nurs. 2016 Aug;12(8):328-335. doi: 10.1016/j.ecns.2016.03.006. No abstract available. PMID 27239244
- [Background] Polivka BJ, Anderson S, Lavender SA, Sommerich CM, Stredney DL, Wills CE, Darragh AR. Efficacy and Usability of a Virtual Simulation Training System for Health and Safety Hazards Encountered by Healthcare Workers. Games Health J. 2019 Apr;8(2):121-128. doi: 10.1089/g4h.2018.0068. Epub 2018 Sep 19. PMID 30234397
- [Background] Polivka BJ, Wills CE, Darragh A, Lavender S, Sommerich C, Stredney D. Environmental Health and Safety Hazards Experienced by Home Health Care Providers: A Room-by-Room Analysis. Workplace Health Saf. 2015 Nov;63(11):512-22; quiz 523. doi: 10.1177/2165079915595925. Epub 2015 Aug 12. PMID 26268486
- [Background] Czuba LR, Sommerich CM, Lavender SA. Ergonomic and safety risk factors in home health care: Exploration and assessment of alternative interventions. Work. 2012;42(3):341-53. doi: 10.3233/WOR-2012-1433. PMID 22523032
- [Background] Wills CE, Polivka BJ, Darragh A, Lavender S, Sommerich C, Stredney D. "Making Do" Decisions: How Home Healthcare Personnel Manage Their Exposure to Home Hazards. West J Nurs Res. 2016 Apr;38(4):411-26. doi: 10.1177/0193945915618950. Epub 2015 Dec 14. PMID 26669605

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-02): https://cdn.clinicaltrials.gov/large-docs/08/NCT06974708/Prot_SAP_000.pdf
  • Informed Consent Form (2025-01-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT06974708/ICF_001.pdf